CLINICAL TRIAL: NCT01409759
Title: Perforator Based Interposition Flaps for Sustainable Release of Burn Scar Contracture: a Reliable, Simple and Versatile Technique. A Randomised Controlled Trial.
Brief Title: Perforator Based Interposition Plasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association of Dutch Burn Centres (Other)
Responsible Party: Association of Dutch Burn Centres, Association of Dutch Burn Centres
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10104 and 10110
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Burn Scar Contraction
Keywords: Perforators; Interposition plasty; Contracture release

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perforator based interposion flap (Experimental): In our concept the flap is designed based on a selected perforator and locally available, preferably normal skin adjacent to the burn scar contracture. The flap consists of skin and underlying subcutaneous tissue. Based on the pre-operative defined perforator, the required length and width and the available preferable normal skin, a design for the perforator flap is made.
  Interventions: Procedure: Perforator based interposition flap
- Full thickness graft (Other)
  Interventions: Procedure: Perforator based interposition flap

INTERVENTIONS:
Procedure: Perforator based interposition flap — The flap is designed based on a selected perforator and locally available, preferably normal skin adjacent to the burn scar contracture. The flap consists of skin and underlying subcutaneous tissue. Based on the pre-operative defined perforator, the required length and width and the available preferable normal skin, a design for the perforator flap is made.

SUMMARY:
Objective: to evaluate the perforator based interposition plasty in comparison to the standard technique (full thickness graft) for scar contracture releases.

Study design: A randomised controlled multicentre intervention study.

Study population: Patients, aged 18 years and older, who require surgery for release of a scar contracture, are eligible for this study. In total 50 patients will be recruited with a follow-up of 3 months post-operatively.

Intervention: A release of the contracture will be performed in combination with òr the standard technique (full thickness graft) òr the perforator based interposition plasty.

Main study parameters/endpoints: the main study parameter is the amount of contraction of the flap/graft after three months.

DETAILED DESCRIPTION:
Rationale:

Scar contracture remains a considerable problem for the burned patient. The standard method of treatment is contracture release in combination with the application of a full or split thickness graft to close the defect. Unfortunately, the effectiveness of skin grafts is limited by scar contraction, which often necessitates additional reconstructions. Moreover, parts of the skin graft may be lost due to poor revascularisation or infection.

Since the discovery of perforator vessels, many types of new flaps can be harvested as long as it incorporates a perforator bundle (artery and vein). This flap design based on perforator vessels and local available skin, should lead to an increased flap survival and superior functional outcome. Based on this concept we developed and explored the possibility of an algorithm for treatment by means of a pilot study performed on 22 patients with a scar contracture. Results show a survival of all flaps of 100% and an expansion of the surface area by 16% after a follow up of at least 3 months. However the implications of the use of perforator based flaps for burn surgery by means of a RCT has yet to be determined.

Primary objective:

Is interpositioned skin of superior quality, as represented by less contraction with the use of the perforator based interposition flaps, compared to the gold standard (full thickness grafts), after 3 months, as measured by transparent sheet planimetry?

Secondary objectives:

* Survival of the flap/graft: i.e. measured by the amount of necrosis
* The quality of the scar: elasticity, colour, subjective scar evaluation

Inclusion criteria are:

* Indication for release of burn scar contracture
* Sufficient tissue for a perforator- based interposition flap (preferably normal skin)
* Able to give informed consent

Exclusion criteria are:

* Age < 18 years
* Location: scars on the face and scalp
* Smoking (however, the patient is eligible if smoking is quit > 3 weeks before the operation)
* Psychiatric disorders (if a loss to follow-up is anticipated)
* Language barrier

ELIGIBILITY:
Inclusion Criteria:

* Indication for release of burn scar contracture
* Sufficient tissue for a perforator- based interposition flap (preferably normal skin)
* Able to give informed consent

Exclusion Criteria:

* Age < 18 years
* Location: scars on the face and scalp
* Smoking (however, the patient is eligible if smoking is quit > 3 weeks before the operation)
* Psychiatric disorders (if a loss to follow-up is anticipated)
* Language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Expansion/contraction of the interpositioned skin after 3 months | 3 months
  Is interpositioned skin of superior quality, as represented by less contraction with the use of the perforator based interposition flaps, compared to the gold standard (full thickness grafts), after 3 months, as measured by transparent sheet planimetry?

CONTACTS AND LOCATIONS:
Overall Officials: Paul P M Van Zuijlen, Prof, Principal Investigator — Red Cross Hospital
Locations (3):
- Netherlands (3):
  - Red Cross Hospital, Beverwijk, North Holland
  - Maastad Hospital, Rotterdam, South Holland
  - Martini Hospital, Burns centre, Groningen